CLINICAL TRIAL: NCT00224133
Title: A Multi-Center, Open-Label Evaluation of the Safety of a New Drug in the Treatment of the Signs and Symptoms of Benign Prostatic Hyperplasia
Brief Title: The Evaluation of the Safety of a New Drug for Benign Prostatic Hyperplasia Used for 9 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Gary Hoel, RPh, PhD, Executive Director of Clinical Research, Watson Laboratories, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SI04011
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2010-04-27 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: benign prostatic hyperplasia, alpha blocker
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — silodosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Silodosin (Experimental): Silodosin 8 mg per day with food
  Interventions: Drug: Silodosin

INTERVENTIONS:
Drug: Silodosin — 8 mg daily
  Other Names: Rapaflo

SUMMARY:
A new drug for benign prostatic hyperplasia is used for 9 months to determine its long-term safety.

DETAILED DESCRIPTION:
This will be a multi-center, open-label 40 week investigation in up to 1,200 men with signs and symptoms of benign prostatic hyperplasia. The following procedures are utilized: physical exams, electrocardiograms, clinical laboratory tests, vital signs, the International Prostate Symptom Score, maximum urine flow rate, adverse events, concomitant medications, and compliance.

All subjects had previously participated in a 12-week double-blind placebo controlled trial (NCT000224107 or NCT000224120)

ELIGIBILITY:
Inclusion Criteria:

* Males in good general health and at least 50 years of age, who have completed SI04009 or SI04010.

Exclusion Criteria:

* Medical conditions that would confound the efficacy evaluation.
* Medical conditions in which it would be unsafe to use an alpha-blocker.
* The use of concomitant drugs that would confound the efficacy evaluation.
* The use of concomitant drugs that would be unsafe with this alpha-blocker.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 661 (Actual)
Dates: Start 2005-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hill, Pharm D, RPh, Study Director — Watson Pharmaceuticals
Locations (79):
- United States (79):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Tucson, Arizona
  - Anaheim, California
  - Carmichael, California
  - Culver City, California
  - Fresno, California
  - Irvine, California
  - La Jolla, California
  - Laguna Woods, California
  - Long Beach, California
  - Newport Beach, California
  - San Bernardino, California
  - San Diego, California
  - Tarzana, California
  - Torrance, California
  - Aurora, Colorado
  - Wheat Ridge, Colorado
  - Waterbury, Connecticut
  - Aventura, Florida
  - Clearwater, Florida
  - Coral Gables, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Plantation, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Marietta, Georgia
  - Chicago, Illinois
  - Melrose Park, Illinois
  - Peoria, Illinois
  - Evansville, Indiana
  - Fort Wayne, Indiana
  - Des Moines, Iowa
  - Overland Park, Kansas
  - Greenbelt, Maryland
  - Boston, Massachusetts
  - Saint Joseph, Michigan
  - Edina, Minnesota
  - Jackson, Mississippi
  - Kansas City, Missouri
  - Missoula, Montana
  - Las Vegas, Nevada
  - Lawrenceville, New Jersey
  - Voorhees Township, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Bay Shore, New York
  - Garden City, New York
  - Kingston, New York
  - Manhasset, New York
  - New York, New York
  - Poughkeepsie, New York
  - Staten Island, New York
  - Williamsville, New York
  - Charlotte, North Carolina
  - Concord, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Bethany, Oklahoma
  - Portland, Oregon
  - Lancaster, Pennsylvania
  - Providence, Rhode Island
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Myrtle Beach, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Lakewood, Washington
  - Seattle, Washington
  - Tacoma, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin

REFERENCES:
- [Result] Marks LS, Gittelman MC, Hill LA, Volinn W, Hoel G. Silodosin in the treatment of the signs and symptoms of benign prostatic hyperplasia: a 9-month, open-label extension study. Urology. 2009 Dec;74(6):1318-22. doi: 10.1016/j.urology.2009.06.072. Epub 2009 Oct 7. PMID 19815265
- See also: FDA approval summary and product label — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.DrugDetails

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 8 mg Silodosin Per Day With Food
Started | 661
Completed | 435
Not Completed | 226
Not completed — Adverse Event | 93
Not completed — Protocol Violation | 6
Not completed — Withdrawal by Subject | 33
Not completed — Lack of Efficacy | 58
Not completed — Lost to Follow-up | 21
Not completed — Physician Decision | 1
Not completed — Other | 14

BASELINE CHARACTERISTICS:
Arm/Group | 8 mg Silodosin Per Day With Food
Number analyzed (Participants) | 661
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 356
  >=65 years | 305
Age Continuous [Mean (Standard Deviation); unit: years] | 65.0 (7.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 661
Region of Enrollment [Number; unit: participants]
  United States | 661

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: All reported adverse events were recorded. Clinically significant abnormal laboratory values or other clinical findings upon examination were also recorded as adverse events.
Time Frame: 9 months
Population: Safety population was analyzed. This population is defined as all enrolled patients who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | 8 mg Silodosin Per Day With Food
Number analyzed (Participants) | 661
participants
  Patients with at least 1 adverse event | 431
  Patients with drug related adverse event | 188
  Patients with a serious adverse events | 29
  Patients with a drug related serious adverse event | 0
  Patients discontinued due to an adverse event | 86
  Discontinued for drug related adverse event | 54

2. Secondary Outcome: International Prostate Symptom Score (IPSS)
Description: The IPSS is a symptom severity scale from 0 to 35 that is derived from a 7 item questionnaire. 0 indicates no symptoms and 35 indicates most severe symptoms.
Time Frame: 9 months
Reporting Status: Not Posted, anticipated posting 2010-03
Measure: Mean (Standard Deviation); unit: Units on a scale

ADVERSE EVENTS:
Time Frame: 9 months
Description: No subject experienced a serious adverse event that was related to treatment.
Arm/Group | 8 mg Silodosin Per Day With Food
Serious Adverse Events (participants affected / at risk) | 29/661
Other Adverse Events (participants affected / at risk) | 138/661
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 mg Silodosin Per Day With Food (N=661)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1)
Arrythmia (Cardiac disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Back injury (Injury, poisoning and procedural complications) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2)
Femoral artery occlusion (Vascular disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 2 (2)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Myocardial infarction (Cardiac disorders) | 1 (1)
Nerve root lesion (Nervous system disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Spinal laminectomy (Surgical and medical procedures) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 mg Silodosin Per Day With Food (N=661)
Retrograde ejaculation (Reproductive system and breast disorders) | 138 (139)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less